CLINICAL TRIAL: NCT01349010
Title: A Randomized, Double Blind, Placebo Control, Multi-center Clinical Study to Evaluate the Efficacy and Safety of Imported Probucol in Hyperlipidemia Patients
Brief Title: Efficacy and Safety of Imported Probucol to Treat Hyperlipidemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Beijing Research Institute (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 009-10-802-01
Record Dates: First submitted 2011-03-24; First posted 2011-05-06 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Hyperlipidemia
Keywords: hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias | interventions — Probucol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo Arm: Placebo 1 tablet bid. p.o
  Interventions: Drug: Placebo
- Probucol (Active Comparator): Probucol Arm: Imported Probucol 250 mg (1 tablet) bid. p.o
  Interventions: Drug: Probucol

INTERVENTIONS:
Drug: Probucol — 250mg (1 tablet) bid. p.o for 8 weeks
  Other Names: Lorelco
  Arms: Probucol
Drug: Placebo — 1 tablet bid. p.o for 8 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of imported Probucol in hyperlipidemia patients.

DETAILED DESCRIPTION:
This is a randomized, double blind, placebo control, multi-centre clinical study in hyperlipidemia patients.

Enrolled subjects will be randomized to the treatment group or control group, and receive Probucol or placebo continuously for 8 weeks; Treatment group: Imported Probucol 250 mg (1 tablet) bid. p.o Control group: Placebo 1 tablet bid. p.o

ELIGIBILITY:
Inclusion Criteria:

1. Signing Informed Content Form;
2. Age >= 20 (the age at the time of signing ICF; both gender);
3. hyperlipidemia patients who meet the following criteria:

   * 4.14 mmol/L (160mg/dL) =< LDL-C (Serum low density lipoprotein-cholesterol) < 6 mmol/L (232mg/dL)
   * TG (Serum triglycerides) < 4.5 mmol/L (398mg/dL);
4. Framingham: Coronary Heart Disease 2-year risk probabilities < 10%.

Exclusion Criteria:

1. Subjects who receive antilipemic agents within 1 month prior to the pre-screening period;
2. Subjects who receive Probucol within 6 months prior to the pre-screening period;
3. Coronary Heart Disease subjects;
4. Subjects being treated with cyclosporine;
5. Subjects with a history of hypersensitivity to Probucol;
6. QTc interval > 450ms (male); QTc interval > 470ms (female);
7. Subjects with impaired hepatic and renal function, who meet any of the following abnormal value:

   * AST >= 100IU/L
   * ALT >= 100IU/L
   * Serum creatinine >= 1.5mg/dL
8. Female subjects who are pregnant, lactating, or who plan to conceive;
9. Subjects who are considered by the investigator to be inappropriate to participate in this trial.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2011-04; Primary Completion 2012-07 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
TC and LDL-C | 8-week
  Changes of TC and LDL-C from the baseline after 8-week treatment;

SECONDARY OUTCOMES:
oxLDL and MCP-1 | 8-week
  Changes of oxLDL and MCP-1 from the baseline after 8-week treatment;

CONTACTS AND LOCATIONS:
Overall Officials: Shuiping Zhao, MD, Principal Investigator — The Sencond Xiangya Hospital of Central South University
Locations (1):
- The Sencond Xiangya Hospital of Central South University, Changsha, Hunan, China